CLINICAL TRIAL: NCT03798379
Title: The Effect of Therapeutic Exercises on Balance, Quality of Life and Pain in Patients Who Were Receiving Neurotoxic Chemotherapy
Brief Title: Exercises for Patients Who Were Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Yeliz Bahar Ozdemir, Principal investigator, Hitit University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2015.278
Record Dates: First submitted 2019-01-04; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: cancer; chemotherapy; peripheral neuropathy; exercise
MeSH Terms: conditions — Neoplasms; Peripheral Nervous System Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Non randomized, single blind, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Active Comparator): Eligible patients who were planned to receive neurotoxic chemotherapy
  Interventions: Other: Exercise
- Control group (No Intervention): Patients eligible for the study and received the 3rd cycle of chemotherapy

INTERVENTIONS:
Other: Exercise — Strengthening, balance and aerobic exercises were explained to the patients examined before chemotherapy sessions and demonstrated by applying on the patient.
  Arms: Exercise group

SUMMARY:
To evaluate the effect of lower extremity strengthening and balance exercises on balance, quality of life and neuropathic pain of the cancer patients receiving neurotoxic chemotherapy.

DETAILED DESCRIPTION:
Cancer-related mortality rates decreased considerably thanks to novel treatment methods and new agents over the last two decades. Although chemotherapy (CT) is an effective treatment type in reducing the size of the tumor and eliminating metastases, it may harm many different organs and systems due to short & long-term side effects. Peripheral neuropathy (PN) is regarded as a neurological and clinical side effect for cancer patients. PN may arise as a paraneoplastic symptom but more commonly occurs with neurotoxic CT agents. Short & long-term side effects that may damage sensory, motor, and autonomic neurons. This damage to the small-fiber sensory nerves causes a change in the sense of touch, pain, and warmth, while the damage to the large-fiber nerves causes a change in the sense of vibration and proprioception. Motor nerve damage affects voluntary movement, muscle tone, and coordination, and damage to the autonomic nervous system affects intestinal motility and blood pressure over smooth muscles. Despite the fact that studies on PN treatment have generally focused on pharmacological agents reducing pain or treating selected side effects, no agent that may be preventive for chemotherapy induced Peripheral Neuropathy (CIPN) due to neurotoxic chemotherapy has been recommended in the review of the American Society of Clinical Oncology.

Side effects due to CT such as anorexia, nausea, vomiting, mucositis, diarrhea, anemia or PN may lead to impairment in the quality of life of the patient and may significantly reduce the level of physical activity. Neurotoxic and ototoxic effects may cause ataxia, paresthesia and dysesthesia, leading to gait, and balance disorders. CIPN has been associated with balance disorder, loss of function and reduced quality of life in the literature. It may result in loss of balance, difficulty in ambulation, increase in the frequency of collapse and accordingly increase in injuries. Despite the fact that medical treatments used in CIPN are often helpful in the treatment of neuropathic pain, no effect has been observed on muscle strength, gait, and balance. It is believed that muscle strength and balance exercises, such as aerobic exercises, can provide mitochondria with oxygen and glucose by increasing blood supply, thereby contributing to energy production and reducing symptoms. Current data suggest that exercise is applicable, safe, and beneficial for this group of patients. Balance exercises at an early stage may prevent or delay the onset of sensory and motor symptoms. Although exercise is accepted as a supportive treatment, which should be addressed more seriously for a patient population with PN, there is not enough information in the literature on timing, frequency, and mode of administration of the treatment program that will be carried out in this specific group of patients.

The aim of this study is to investigate the effects of therapeutic exercise program including concurrently initiated strengthening, balance and aerobic exercises on the symptoms, balance status and quality of life of the group of patients who have a limited physical activity, a risk of developing PN following the treatment, and will have a long-term bed rest and compare with the group of patients not receiving any exercise program in the same treatment period.

ELIGIBILITY:
Inclusion Criteria:

* the ability to understand the informed consent form, and the signing the informed consent form after being informed in detail,
* planned to have ≥3 cycles of neurotoxic chemotherapy (paclitaxel, docetaxel from taxane class agents, and cisplatin, oxaliplatin or carboplatin from platin group),
* expected to have a survival of ≥6 months,
* to have an Eastern Cooperative Oncology Group performance level between 0-2,
* to have a full manual muscle strength.

Exclusion Criteria:

* Previously diagnosed peripheral neuropathy (Diabetic peripheral neuropathy, entrapment neuropathies etc.)
* Patients receiving medical treatment due to neuropathic pain (pregabalin, gabapentin, duloxetine etc.)
* Pre-existing neurological disease
* Pre-existing diabetes mellitus (>3 years or insulin use)
* Alcoholism
* HIV infection
* Presence of peripheral vascular disease
* Vitamin D or vitamin B12 deficiency
* Non-ambulatory or refuse to practice exercise program
* Visual or vestibular system impairment
* Patients with central nervous system involvement or metastasis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Balance assessment | 3 months
  NeuroCom Balance Master® device (Natus Medical, San Carlos, California, USA) is a balance evaluation device measuring the position of the center of gravity, postural control along with static and dynamic stability.

SECONDARY OUTCOMES:
Berg balance scale | 3 months
  Berg balance scale used in the evaluation of balance based on performance is a 14-item measure in which patient is required to perform different activities.14 different activities are scored between 0 (worst) and 4 (best) according to the patient's performance. The maximum score is 56. A total score close to 56 indicates that the balance of patient is good.
PainDETECT: questionnaire | 3 months
  The presence of neuropathic pain was evaluated with the painDETECT questionnaire. The maximum score is 35 and a high score indicates the severity of neuropathic pain. When the PD-Q score is more than 13, it is indicated the presence of neuropathic pain component.
The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire | 3 months
  It is a questionnaire developed by the European Organization for Research and Treatment of Cancer and used to assess the quality of life of cancer patients participating in clinical trials and includes a variety of components. Patients' higher points of functional scale and general health status scale and lower points of symptom scale scores indicate a high QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zimmer P, Trebing S, Timmers-Trebing U, Schenk A, Paust R, Bloch W, Rudolph R, Streckmann F, Baumann FT. Eight-week, multimodal exercise counteracts a progress of chemotherapy-induced peripheral neuropathy and improves balance and strength in metastasized colorectal cancer patients: a randomized controlled trial. Support Care Cancer. 2018 Feb;26(2):615-624. doi: 10.1007/s00520-017-3875-5. Epub 2017 Sep 30. PMID 28963591
- [Background] Streckmann F, Kneis S, Leifert JA, Baumann FT, Kleber M, Ihorst G, Herich L, Grussinger V, Gollhofer A, Bertz H. Exercise program improves therapy-related side-effects and quality of life in lymphoma patients undergoing therapy. Ann Oncol. 2014 Feb;25(2):493-9. doi: 10.1093/annonc/mdt568. PMID 24478323
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Cammisuli S, Cavazzi E, Baldissarro E, Leandri M. Rehabilitation of balance disturbances due to chemotherapy-induced peripheral neuropathy: a pilot study. Eur J Phys Rehabil Med. 2016 Aug;52(4):479-88. Epub 2016 May 31. PMID 27243828
- [Background] Nurgalieva Z, Xia R, Liu CC, Burau K, Hardy D, Du XL. Risk of chemotherapy-induced peripheral neuropathy in large population-based cohorts of elderly patients with breast, ovarian, and lung cancer. Am J Ther. 2010 Mar-Apr;17(2):148-58. doi: 10.1097/MJT.0b013e3181a3e50b. PMID 19417586
- [Background] Hershman DL, Lacchetti C, Loprinzi CL. Prevention and Management of Chemotherapy-Induced Peripheral Neuropathy in Survivors of Adult Cancers: American Society of Clinical Oncology Clinical Practice Guideline Summary. J Oncol Pract. 2014 Nov;10(6):e421-e424. doi: 10.1200/JOP.2014.001776. No abstract available. PMID 29424607